CLINICAL TRIAL: NCT05076890
Title: Hemp 15 mg & 50 mg Capsule Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia Herbs Inc. (Industry)
Collaborators: Appalachian College of Pharmacy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Gaia-19002
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-08

CONDITIONS: Absorption; Chemicals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 mg/g Full Spectrum Hemp Extract (Experimental): A single capsule of 15 mg/g Full Spectrum Hemp Extract will be delivered.
  Interventions: Dietary Supplement: 15 mg/g Full Spectrum Hemp Extract
- 50 mg/g Full Spectrum Hemp Extract (Experimental): A single capsule of 50 mg/g Full Spectrum Hemp Extract will be delivered.
  Interventions: Dietary Supplement: 50 mg/g Full Spectrum Hemp Extract

INTERVENTIONS:
Dietary Supplement: 15 mg/g Full Spectrum Hemp Extract — HPMC capsules containing full spectrum standardized hemp extract in liquid form.
  Arms: 15 mg/g Full Spectrum Hemp Extract
Dietary Supplement: 50 mg/g Full Spectrum Hemp Extract — HPMC capsules containing full spectrum standardized hemp extract in liquid form.
  Arms: 50 mg/g Full Spectrum Hemp Extract

SUMMARY:
This study is intended to investigate the absorption of cannabidiol (CBD) and cannabidiol acid (CBD-A) in plasma from an oral delivery of a single dose of full spectrum hemp extract at two concentrations over a 4-hour timeline.

DETAILED DESCRIPTION:
This study is designed to determine the time to maximum plasma concentration of CBD and CBD-A after an oral dose of standardized full spectrum hemp extract over a 4-hour timeline. This study is designed to include two arms. Each arm will be delivered a different concentration of standardized full spectrum hemp extract, either 15 mg or 50 mg. Throughout the course of the study all participants will be asked to provide four (4) plasma samples, 10 randomly selected participants will be asked to provide five (5) plasma samples. Samples will then be evaluated using a validated LC-MS/MS method to develop a blood concentration time curve in order to determine time to reach maximum blood concentration. This trial is double-blinded with two arms enrolling only healthy individuals. The participants randomized for a fifth blood draw will be randomly selected from these two arms.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Ages 18 - 65.
4. In good general health as evidenced by medical history as indicated by oral confirmation of study participant.
5. Ability and willingness to suspend the use of any other herbal dietary supplements for 48 hours prior the first clinical visit associated with this study.
6. Ability and willingness to abstain from alcohol use for 12 hours prior to the first clinical visit.
7. Cannabis and CBD naïve for 60 days or more prior to enrolling in the study.
8. Ability and willingness to abstain from food for 6 hours prior to the first clinical visit.

Exclusion Criteria:

1. Current use of regular medication for a chronic condition.
2. Current pregnancy or lactation.
3. Plans to become pregnant during the intended duration of the study.
4. Known allergic reactions to hemp flower.
5. Known severe food allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Time to maximum plasma concentration | Over 4 hours
  To determine the time to maximum plasma concentration of cannabidiol (CBD) and cannabidiol acid (CBD-A) from an oral delivery of a single dose of standardized 15 mg or 50 mg full spectrum hemp extract

SECONDARY OUTCOMES:
Detectable THC | Over 4 hours
  To determine if the oral delivery of a full spectrum hemp extract standardized to less than 0.3% ∆^9- tetrahydrocannabinol (THC) results in detectable amounts of THC in plasma.

OTHER OUTCOMES:
Present in measurable amount over time | 7 - 10 days
  To determine if CBD, CBD-A, or THC are present 7 to 10 days after a single oral dose of 15 mg or 50 mg standardized full spectrum hemp extract.

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian College of Pharmacy, Oakwood, Virginia, United States

IPD SHARING:
Plan to Share IPD: No